CLINICAL TRIAL: NCT03599024
Title: Patient-controlled Epidural Analgesia Versus Conventional Epidural Analgesia After Total Hip Replacement - a Randomized Trial
Brief Title: Role of Patient-controlled Epidural Analgesia After Total Hip Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Ostrava (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FNO-KARIM-07-PCEA; MH CZ - DRO-FNOs/2014 (Other Grant/Funding Number: Ministry of Health of the Czech Republic)
Record Dates: First submitted 2018-05-16; First posted 2018-07-26 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Hip Joint Disorders
Keywords: patient-controlled analgesia; epidural analgesia; analgesics; drug consumption; total hip replacement; pain relief
MeSH Terms: interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Intervention Model Description: The patients were randomized into two groups with two distinct interventions - patient-controlled analgesia vs. conventional analgesia prescribed by the attending physician.
Masking Description: Neither the investigators nor the patients were blinded in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PCEA Group (Experimental): The patients randomized into this arm were able to control the administration of analgesics, according to their subjective condition.
  Interventions: Procedure: PCEA; Procedure: Total hip replacement
- Non-PCEA Group (Active Comparator): The patients randomized into this arm were receiving analgesics according to the physician's prescription.
  Interventions: Procedure: Non-PCEA; Procedure: Total hip replacement

INTERVENTIONS:
Procedure: PCEA — The patients were able to control the administration of analgesics by themselves.
  Other Names: Patient-controlled epidural analgesia (PCEA)
  Arms: PCEA Group
Procedure: Non-PCEA — The patients were receiving analgesics according to the physician's prescription.
  Other Names: Non-patient controlled epidural analgesia (Non-PCEA)
  Arms: Non-PCEA Group
Procedure: Total hip replacement — All patients enrolled in the study were indicated for total hip replacement surgery.

SUMMARY:
Total hip replacement (THR) is frequently followed by high pain experience. Epidural analgesia is a mainstay in postoperative treatment in patients after THR. The investigators found that patient-controlled epidural analgesia (PCEA) decreases total analgesics consumption compared to conventional method of analgesia based on physician's prescription while maintaining similar pain relief and safety profile. Therefore, PCEA should be considered the first choice method of analgesia in patients undergoing THR.

DETAILED DESCRIPTION:
The prospective, randomized controlled trial was performed at University Hospital Ostrava. All eligible participants were adult patients of both genders aged 18 years or older, and scheduled for elective orthopaedic surgery (THR). The enrolled patients underwent per-protocol randomization into one of two groups (PCEA or non-PCEA group) using the envelopes method. Randomization was performed immediately after ICU admission by an independent physician, who was not involved in the data collection or management of the study subjects. Following randomization, patients were admitted to the ICU. Data for the analyses were collected for 24 hours after THR. The baseline demographic and preoperative characteristics (age, gender, weight, body mass index, and American Society of Anesthesiologists [ASA] physical status) were obtained at the time of admission. The degree of motor block was assessed using the modified Bromage Score. The level of sedation due to the residual effect of anaesthetics at the time of admission was assessed using a sedation score. The Visual Analogue Scale (VAS) values were determined at hourly intervals and 30 minutes after administration of analgesics to determine the effect of the analgesic dose. The other parameters evaluated at hourly intervals were: a) the presence of hypotension defined as a decrease in systolic blood pressure below 90 mmHg or a greater than 30% decrease from the baseline value; b) bradypnea measured on a numeric scale; c) bradycardia defined as heart rate ≤ 50/min and tachycardia defined as heart rate ≥ 120/min; d) the presence of postoperative nausea and vomiting (PONV); and e) skin itching. At the time of discharge from the ICU, the total consumption of analgesics was recorded, and patients' satisfaction was evaluated using the Likert scale. All patients were perioperatively treated by the protocol for administration of anesthesia and analgesia: The patients were administered 7.5 mg of midazolam orally one hour before surgery. Patients weighing more than 70 kg received 2 mg of bisulepin. Prior to surgery, a subarachnoid blockade was established with 2-4 ml of levobupivacaine 0.5% at the L2-L3 spinal interspace. Subsequently, a catheter for postoperative analgesia was inserted into the epidural space. If the subarachnoid blockade was insufficient for surgery, epidural levobupivacaine 0.5 % was administered to a maximum dose of 10 ml, after which the patient underwent general anesthesia and was excluded from the study. During surgery, patients were sedated with a target-controlled infusion of propofol (dose of 1-2 mg/kg body weight per hour) so that they were asleep but aroused when spoken to. After surgery, patients received a mixture of levobupivacaine 0.1% and sufentanil 1 µg/ml. Postoperatively, patients were moved to the ICU. Immediately after ICU admission, continuous monitoring of vital functions and pain was initiated. When the pain intensity exceeded ≥ 4 points, analgesic therapy was initiated by the administration of a mixture containing levobupivacaine 0.1% and sufentanil 1 μg/ml. The PCEA group was initially given a bolus of 10 ml of the mixture, and then a basal infusion at the rate of 3 ml/h. The bolus was set on 4 ml, a lockout interval of 20 minutes, and a maximum dose of 40 ml/4 h according to the literature recommendation. The non-PCEA group was initially administered 5 ml of the analgesic mixture followed by a basal infusion at 5 ml/h. If pain developed, a bolus of 8 ml of the mixture was administered according to the physician's prescription. If analgesia was insufficient after 1 hour of maximal dosing in both groups, the patient was given adjunctive analgesic therapy including one or a combination of the following drugs: i.v. paracetamol, i.v. metamizole, or i.v. tramadol. Patients requiring systemic adjunctive medication were excluded from the final analysis.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* ASA I-III on pre-anesthesia evaluation
* ICU admission after total hip replacement surgery
* Glasgow Coma Scale (GCS) 13 or more
* Spontaneous breathing at a rate of 12-24 breaths/min
* SpO2 ≥ 90%
* Modified Bromage Score 0 or 1
* Visual analog scale (VAS) ≥ 4
* Signed Informed Consent Form for participation

Exclusion Criteria:

* History of long-term opioid therapy (the use of an opioid analgesic at doses higher than codeine 120 mg/day, hydrocodone 40 mg/day, tramadol 200 mg/day or oxycodone 40 mg/day 0-4 days before surgery)
* Indications for revision surgery during immediate postoperative care
* Acute skin disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2014-09-01 (Actual); Primary Completion 2015-12-01 (Actual); Study Completion 2016-03-31 (Actual)

PRIMARY OUTCOMES:
Difference in consumption of analgesics | 18 months
  The primary goal of this prospective, randomized study was to compare the effects of two different sufentanil-based methods of analgesia; patient controlled (PCEA) and conventional non-PCEA) where drug is delivered according to the physician's prescription. The main goal was to determine any difference in total consumption of analgesics.

SECONDARY OUTCOMES:
Patient satisfaction - 24 hours after surgery | 24 hours
  Patient satisfaction was assessed using the Likert scale for the period of 24 hours after surgery.
Degree of pain intensity - 24 hours after surgery | 24 hours
  The degree of pain intensity was assessed in patients in both groups. The Visual Analogue Scale (VAS) values were determined at hourly intervals and 30 minutes after administration of analgesics to determine the effect of the analgesic dose. A Visual Analogue Scale (VAS) is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured.
Safety of analgesics administration - hypotension | 24 hours
  The safety of the methods of analgesia based on the occurrence of analgesia-related complications measured with the presence of hypotension defined as a decrease in systolic blood pressure below 90 mmHg or a greater than 30% decrease from the baseline value.
Safety of analgesics administration - bradypnea | 24 hours
  The safety of the methods of analgesia based on the occurrence of analgesia-related complications measured with the presence of bradypnea measured on a numeric scale: (1= normal respiratory rate [RR]; 2 = RR ≤ 12/min; and 3 = RR ≤ 8/min)
Safety of analgesics administration - heart rate abnormalities | 24 hours
  The safety of the methods of analgesia based on the occurrence of analgesia-related complications measured with the presence of bradycardia defined as heart rate ≤ 50/min and tachycardia defined as heart rate ≥ 120/min.
Safety of analgesics administration - PONV | 24 hours
  The safety of the methods of analgesia based on the occurrence of analgesia-related complications measured with the presence of PONV as determined using a numerical scale (0 = no nausea; 1 = mild nausea; 2 = antiemetic given; 3 = nausea despite antiemetic; and 4 = vomiting)11; and e) skin itching (yes/no).

CONTACTS AND LOCATIONS:
Overall Officials: Renáta Zoubková, PhDr., Principal Investigator — University Hospital Ostrava
Locations (1):
- University Hospital Ostrava, Ostrava, Moravian-Silesian Region, Czechia

IPD SHARING:
Plan to Share IPD: No
The investigators do not plan to share the individual participant data with other researchers.

REFERENCES:
- [Background] Sinatra RS, Torres J, Bustos AM. Pain management after major orthopaedic surgery: current strategies and new concepts. J Am Acad Orthop Surg. 2002 Mar-Apr;10(2):117-29. doi: 10.5435/00124635-200203000-00007. PMID 11929206
- [Background] Singelyn FJ, Ferrant T, Malisse MF, Joris D. Effects of intravenous patient-controlled analgesia with morphine, continuous epidural analgesia, and continuous femoral nerve sheath block on rehabilitation after unilateral total-hip arthroplasty. Reg Anesth Pain Med. 2005 Sep-Oct;30(5):452-7. doi: 10.1016/j.rapm.2005.05.008. PMID 16135349
- [Background] Hartrick CT, Bourne MH, Gargiulo K, Damaraju CV, Vallow S, Hewitt DJ. Fentanyl iontophoretic transdermal system for acute-pain management after orthopedic surgery: a comparative study with morphine intravenous patient-controlled analgesia. Reg Anesth Pain Med. 2006 Nov-Dec;31(6):546-54. doi: 10.1016/j.rapm.2006.08.011. PMID 17138198
- [Background] Bertini L, Mancini S, Di Benedetto P, Ciaschi A, Martini O, Nava S, Tagariello V. Postoperative analgesia by combined continuous infusion and patient-controlled epidural analgesia (PCEA) following hip replacement: ropivacaine versus bupivacaine. Acta Anaesthesiol Scand. 2001 Jul;45(6):782-5. doi: 10.1034/j.1399-6576.2001.045006782.x. PMID 11421841
- See also: Website dealing with post-operative pain management. — https://www.postoppain.org/methodology/